CLINICAL TRIAL: NCT00846404
Title: Markers of Oxidative Stress Present in Blood in Patients With Diastolic Dysfunction
Brief Title: Markers of Oxidative Stress Diastolic Dysfunction
Acronym: ODDS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Emory University (Other)
Responsible Party: Tai-Hwang Michael Fan, MD, PhD, Atlanta VAMC
Other Study IDs: 730-2006
Record Dates: First submitted 2009-02-16; First posted 2009-02-18 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Diastolic Heart Failure; Diastolic Dysfunction
Keywords: heart failure; cardiomyopathy; diastolic dysfunction
MeSH Terms: conditions — Heart Failure, Diastolic; Heart Failure; Cardiomyopathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case: Patients with Diastolic Dysfunction
- Control: Patients without Diastolic Dysfunction

SUMMARY:
This study is to look at the differences between people who have evidence of abnormal heart relaxation (diastolic dysfunction) on sound wave pictures of the heart (an echocardiogram) compared to those who do not. If you have abnormal relaxation, it can be a cause of shortness of breath or can be present without knowing about it.

A condition known as oxidative stress mayb e associated with this abnormal relaxation. This condition occurs when abnormal oxygen injures heart cells. We would like to learn if patients with abnormal relaxation have increased oxidative stress.

DETAILED DESCRIPTION:
Background

Introduction:

The incidence of congestive heart failure (CHF) has been increasing significantly. Between 1971 and 1994, the crude hospitalization rate for heart failure increased from 8.2 to 33.8 per 1000 suggesting a marked rise in the prevalence of this condition.1,2 Furthermore, data from the Framingham study suggest that the incidence of CHF doubles with each advancing decade of age after 45.2 About 43% of individuals with CHF have normal systolic function, or diastolic heart failure.3 The occurrence of diastolic heart failure is more frequent in women and individuals with hypertension, coronary artery disease, obesity, and diabetes mellitus and is associated with a significant increase in mortality.

Diastolic heart failure and diastolic dysfunction are common disorders, characterized by delayed ventricular relaxation and increased diastolic stiffness in the absence of systolic dysfunction. Nitric oxide (NO•) may contribute to the pathophysiology of these disorders as well as many other processes. In peripheral tissue, NO is a potent vasodilator produced by endothelial cells and is thought to mediate vascular relaxation in response to acetylcholine, bradykinin, and substance P. In multiple animal model studies, endothelial production of NO• has disproportionately enhances diastolic left ventricular function without a substantial effect on early systolic pressure development. This was shown in ferret papillary muscles in response to Substance P and recapitulated in mouse models using a cGMP analogue as a surrogate for NO•.

Both diastolic dysfunction and diastolic heart failure are intimately related to hypertension. Recently, we have observed increased oxidative stress and decreased NO• availability in a mouse model that develop diastolic dysfunction. Specifically, in a deoxycorticosterone-induced hypertensive mouse, in which diastolic dysfunction develops, there is evidence of endothelial nitric oxide synthase (eNOS) dysfunction that can be prevented by addition of a reduced cofactor, tetrahydrobiopterin (BH4). It is well known that hypertension is associated with increased oxidative stress and BH4 oxidation. When BH4 is oxidized, eNOS ceases to make NO•. We believe that when this happens in the myocardium, the lack of cardiac NO• results in diastolic dysfunction that will be treatable with BH4 supplementation. A corollary of this hypothesis is that humans with diastolic dysfunction will be more oxidized than those case matched controls without diastolic dysfunction (figure 1).

There are several ways to measure oxidative stress in humans. Among the most convenient and least invasive are to measure lipid peroxides (derivatives of reactive oxygen metabolites, dROMs), isoprostanes, and oxidized and reduced glutathione ratios. Glutathione is an important water-phase antioxidant and essential cofactor for antioxidant enzymes. It provides protection endogenous oxygen radicals. Since glutathione can exist in oxidized and reduced forms, it can serve as a buffer for increased oxidative stress. Moreover, the relative amounts of these two forms are a reflection of the oxidative state of humans. Recently, we have submitted a manuscript showing that we can effectively measure oxidative stress out of the blood of patients and that this measure differentiates between people with an without atrial fibrillation, an abnormal heart beat for which there is growing evidence that oxidative stress plays a role.

Objectives:

Based on the discussion above, we hypothesize that patients with diastolic dysfunction will show higher levels of blood oxidative stress than a case matched control group. This will be tested by comparing oxidative stress markers from the blood of patients with and without diastolic dysfunction. The study design will be a case-control format with controls matched for age (by decade), smoking, and diabetes. If the hypothesis is true, it could lead to new, more effective treatments for cardiac diastolic dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Patients age ≥ 18 years.
* Able to provide informed consent.
* Cases must have diastolic dysfunction documented by echocardiography an interval of six month before the time of enrollment.

Exclusion Criteria:

* Control subjects must not have diastolic dysfunction documented by echocardiography in an interval of six month before the time of enrollment.
* All subjects will be in sinus rhythm.
* All patients will have a left ventricular ejection fraction of > 55% but less than < 70%.
* All patients will have normal systolic and diastolic cardiac dimensions on the qualifying echocardiogram.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of primary care cardiology clinics at Emory University.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2006-07; Primary Completion 2007-05 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Evidence of diastolic dysfuntion documented by echocardiography with six months before the time of enrollment. | Documented six month before the time of enrollment.

SECONDARY OUTCOMES:
This study is observational. It entails measurement products from a blood draw. | One visit that is at enrollment. No follow ups.

CONTACTS AND LOCATIONS:
Overall Officials: Tai-Hwang M Fan, MD, PhD, Principal Investigator — Emory Univeristy IRB
Locations (1):
- Atlanta VAMC, Decatur, Georgia, United States